CLINICAL TRIAL: NCT00955981
Title: Randomized, Double-Blind, Multicenter, Placebo-Controlled, Safety and Efficacy Study of RDEA594 Versus Placebo in the Treatment of Hyperuricemia in Patients With Gout
Brief Title: Gout Dose Response Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDEA594-202
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — lesinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- RDEA594 200 mg qd for 28 days (Experimental)
  Interventions: Drug: RDEA594
- RDEA594 200 mg, 400 mg (Experimental): RDEA594 200 mg qd for 7 days followed by 400 mg qd for 21 days
  Interventions: Drug: RDEA594
- RDEA594 200 mg, 400 mg and 600 mg (Experimental): RDEA594 200 mg qd for 7 days followed by 400 mg qd for 7 days followed by 600 mg qd for 14 days
  Interventions: Drug: RDEA594
- Matching placebo (Placebo Comparator): RDEA594 matching placebo qd for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDEA594 — Uricosuric agent for the treatment of gout
  Arms: RDEA594 200 mg qd for 28 days; RDEA594 200 mg, 400 mg; RDEA594 200 mg, 400 mg and 600 mg
Drug: Placebo — Matching placebo
  Arms: Matching placebo

SUMMARY:
To compare the proportion of subjects whose serum urate (sUA) level is < 6.0 mg/dL after 28 days of dosing by treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Male or post-menopausal or surgically sterile female.
* 18 - 75 years of age.
* Hyperuricemic (i.e., screening sUA ≥8 mg/dL).
* Meets criteria for the diagnosis of gout as per the American Rheumatism Association (ARA) Criteria for the Classification of Acute Arthritis of Primary Gout.
* Willing and able to give informed consent and adhere to visit/protocol schedules (informed consent must be given before the first study procedure is performed).
* Subjects entering the optional Extension Period must have successfully completed the Double-Blind Treatment Period and Follow-up Period within approximately 4 months and must not have experienced any serious adverse events considered possibly related to study drug.

Exclusion Criteria:

* Classified as an overproducer of urine urate (Cur > 6.0 ml/min/1.73 m2 24- hour urine).
* Consumes more than 14 drinks of alcohol per week (e.g., 1 drink = 5 oz [150 ml] of wine, 12 oz [360 ml] of beer, or 1.5 oz [45 ml] of hard liquor).
* History or suspicion of drug abuse.
* Documented history of or suspicion of kidney stones.
* History of rheumatoid arthritis or other autoimmune disease.
* Confirmed (positive serology to HIV1 and HIV 2) or suspected HIV infection.
* Positive serology to HCV antibodies (Abs), and/or hepatitis B surface antigen (HBsAg).
* History of malignancy, except treated non-melanomatous skin cancer or cervical dysplasia.
* History of cardiac abnormalities, including abnormal and clinically relevant ECG changes such as bradycardia (sinus rate <45 bpm), complete left bundle branch block (LBBB), second or third degree heart block, intraventricular conduction delay with QRS duration >120 msec, symptomatic or asymptomatic arrhythmias with the exception of sinus arrhythmia, evidence of ventricular pre-excitation, frequent palpitations or syncopal episodes, heart failure, hypokalemia, family history of Long QT Syndrome, and/or family history of sudden death in an otherwise healthy individual between the ages of 1 and 30 years.
* Any condition predisposing them to QT prolongation including pathological Q-wave (defined as Q-wave >40 msec or depth > 0.4-0.5 mV).
* Any use of a concomitant medication that prolong the QT/QTc interval within the 14 days prior to Baseline (Day 0)
* QT interval corrected for heart rate according to Fridericia (QTcF) > 450 msec at Screening or pre-dose at Baseline (Day 0)
* Uncontrolled hypertension (above 150/95)
* Inadequate renal function
* Hemoglobin < 10 g/dL (males) or < 9 g/dL (females)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN)
* Gamma glutamyl transferase (GGT) > 3 x ULN
* Active peptic ulcer disease requiring treatment
* History of xanthinuria, active liver disease, or hepatic dysfunction.
* Requires therapy with any other urate-lowering medication, other than the study medication.
* Requires long-term use of salicylates; diuretics; azathioprine; mercaptopurine; theophylline; intravenous colchicine; cyclosporine; cyclophosphamide; pyrazinamide; sulfamethoxazole; or trimethoprim
* Taking medications known as enzyme inducers
* Receiving a strong or moderate inhibitor of CYP3A4 or a P-gp inhibitor within 1 month prior to study drug dosing
* Gout flare at screening that is resolved for less than one week prior to the first treatment with study medication (exclusive of chronic synovitis/ arthritis)
* Female of childbearing potential
* Received an investigational medication within 4 weeks prior to study medication administration
* Previously participated in a clinical study involving RDEA806 or RDEA594.
* Known hypersensitivity or allergy to RDEA594 or colchicine or any components in their formulations.
* Body mass index (BMI) >40 kg/m2.
* Taking greater than 1000 mg/day of Vitamin C.
* Any other medical or psychological condition, which in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.
* Inadequate renal function after completing the Double-Blind Treatment period prior to entering Extension Period.
* Requiring treatment with prohibited medications noted in exclusion criteria numbers 20-23 after completing the Double-Blind Treatment Period prior to entering the Extension Period.
* Clinically relevant medical event as determined by the investigator in consultation with medical monitor prior to entering the Extension Period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To compare the proportion of subjects whose serum urate (sUA) level is < 6.0 mg/dL after 28 days of dosing by treatment group. | 28 Days

SECONDARY OUTCOMES:
To evaluate the proportion of subjects whose sUA levels are <6.0 mg/dL, <5.0 mg/dL and <4.0 mg/dL at each weekly study visit during the Double-Blind Period. | 28 Days
To evaluate the absolute and percent reduction from baseline in sUA levels at each weekly study visit. | 28 Days and through extension
To evaluate the percentage change in 24-hour urine urate level (excretion) from baseline to Day 28. | 28 Days and through extension
To evaluate the incidence of gout flares. | 28 Days and through extension
To evaluate the safety and tolerability of RDEA594 in subjects with gout. | 28 Days and through extension
To evaluate the proportion of subjects whose sUA level decreases to or is maintained at <6.0 mg/dL in the Open-Label Extension Period. | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Hingorani, MD, PhD, MBA, Study Director — Ardea Biosciences, Inc.
Locations (26):
- United States (4):
  - Los Angeles, California
  - DeLand, Florida
  - Winston-Salem, North Carolina
  - Jackson, Tennessee
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Plovidv
  - Sofia
  - Varna
- Canada (5):
  - Coquitlam, British Columbia
  - Kelowna, British Columbia
  - Thornhill, Ontario
  - Toronto, Ontario
  - Mirabel, Quebec
- Czechia (2):
  - Bruntál
  - Prague
- Tbilisi, Georgia
- Germany (3):
  - Goch
  - Hamburg
  - Nuremberg
- Poland (6):
  - Elblag
  - Lodz
  - Lublin
  - Poznan
  - Radom
  - Wroclaw